CLINICAL TRIAL: NCT05582525
Title: Relationship Between the Coronavirus 2019 Disease (COVID-19) Vaccines and the Development of New Lower Urinary Tract Symptoms: A Cross-sectional Study on Medical Students.
Brief Title: COVID-19 Vaccines and the Development of New LUTS
Status: Completed | Type: Observational
Sponsor: The Hashemite University (Other)
Responsible Party: Principal Investigator, Jad Khaled AlSmadi, Urology Clinic, The Hashemite University
Other Study IDs: 24/6/2021/2022
Record Dates: First submitted 2022-10-14; First posted 2022-10-17 (Actual); Last update posted 2022-10-17 (Actual); Status verified 2022-10

CONDITIONS: COVID-19 Vaccine Adverse Reaction; Lower Urinary Tract Symptoms
Keywords: COVID-19 Vaccines; LUTS; Medical students
MeSH Terms: conditions — Lower Urinary Tract Symptoms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study was conducted to check whether coronavirus disease 2019 (COVID) vaccines have a relationship with LUTS or not in a healthy and mostly medically free population.

ELIGIBILITY:
Inclusion Criteria:

1. Medical Student
2. Having had a COVID-19 Vaccine

Exclusion Criteria:

None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Medical students
Sampling Method: Non-Probability Sample
Enrollment: 341 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-04-01 (Actual)

PRIMARY OUTCOMES:
New Lower Urinary Tract Symptoms | 2-3 months
  Only after having had any COVID -19 vaccine

CONTACTS AND LOCATIONS:
Overall Officials: Jad K AlSmadi, MD, Principal Investigator — The Hashemite University
Locations (1):
- The Hashemite University, Zarqa, Jordan

IPD SHARING:
Plan to Share IPD: No
The data are going to be kept safe on the internet-based questionnaire website. Only the study team will be able to see those information.